CLINICAL TRIAL: NCT03260439
Title: Doses Tramadol With Bupivacaine in Penial Block Improve Efficiency of Postoperative Analgésia in Children in Circumcision
Brief Title: Tramadol in Penial Block Does it Improve Efficiency of Postoperative Analgesia in Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leila mansali stambouli (Other)
Responsible Party: Sponsor-Investigator, Leila mansali stambouli, Principal Investgator and ClinicalProfessor, University of Monastir
Organization: University of Monastir (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: OMB NO: 0925-0586
Record Dates: First submitted 2017-08-18; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Tramadol - Anesthetics- Child - Circumcision
Keywords: tramadol-penile block -circumcision surgery-anesthesia-child
MeSH Terms: interventions — Tramadol

STUDY DESIGN:
Intervention Model Description: Randomized, controlled and double blind assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G1 (group BT) (Other): The children were randomized to 2 groups (n = 53 in each group) to receive 0.1% BPV non-adrenalinated 0.5% / kg on each side with tramadol 2mg / Kg (G1: GroupBT ). Tramadol
  Interventions: Drug: Tramadol
- G2 (group B or control) (Other): The children were randomized to 2 groups (n = 53 in each group) to receive 0.1% BPV non-adrenalinated 0.5% / kg on each side with saline serum at the same volume (G2: Group B or control). Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tramadol — Children receive 0.1% BPV non-adrenalinated 0.5% / kg on each side with tramadol 2mg / Kg (G1: GroupBT ). Postoperativ analgesia was assessed by: the modified OPS scale at waking (H0), 1st (H1), 2nd (H2), and 24th (H24) PO hour at home, by the number of analgesic The hospital and home, and by the time of the first demand analgesic.
  Other Names: group BT
  Arms: G1 (group BT)
Drug: Placebo — Children receive 0.1% BPV non-adrenalinated 0.5% / kg on each side with saline serum at the same volume (G2: Group B or control). Postoperativ analgesia was assessed by: the modified OPS scale at waking (H0), 1st (H1), 2nd (H2), and 24th (H24) PO hour at home, by the number of analgesic The hospital and home, and by the time of the first demand analgesic.
  Other Names: group B or control
  Arms: G2 (group B or control)

SUMMARY:
After the consent of the local ethics committee and informed consent of the parents, we conducted a prospective randomized, double-blind study, from 30 June 2014 to 31 December 2014, including one to eight year olds, ASA I or II and Programmed for circumcision.We collected 53 children in each group.

DETAILED DESCRIPTION:
After the consent of the local ethics committee and informed consent of the parents, we conducted a prospective randomized, double-blind study, from 30 June 2014 to 31 December 2014, including one to eight year olds, ASA I or II and Programmed for circumcision. Anesthesia was induced with sevoflurane at 8% and maintained by the same agent at 2%. The children were randomized to 2 groups (n = 53 in each group) to receive 0.1% BPV non-adrenalinated 0.5% / kg on each side with either tramadol 2mg / Kg (G1: GroupBT ) Or saline serum at the same volume (G2: Group B or control). Postoperative analgesia was assessed by: the modified OPS scale at waking (H0), 1st (H1), 2nd (H2), and 24th (H24) PO hour at home, by the number of analgesic inThe hospital and at home, and by the time of the first demand analgesic.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II
* Were scheudled to circumcision surgery
* Performed by experenced surgeon under general anesthesia

Exclusion Criteria:

* children with full stomach
* A history of gastric reflux
* A history of cardiovascular or neuromuscular disease
* Allergies to the study drugs

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia | from awake until 60 min after emergence
  Postoperative analgesia was assessed by modified OPS scale, by the number of the
  number of analgesic in The hospital and home, and by the time of the first demand analgesic.

CONTACTS AND LOCATIONS:
Overall Officials: leila Mansali Stambouli, MD PhD, Principal Investigator — University Hospital of Fattouma Bourguiba Monastir TUNISIA
Locations (1):
- University Hospital of Fattouma Bourguiba, Monastir, Monastir- Tunisia, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kargi E, Isikdemir A, Tokgoz H, Erol B, Isikdemir F, Hanci V, Payasli C. Comparison of local anesthetic effects of tramadol with prilocaine during circumcision procedure. Urology. 2010 Mar;75(3):672-5. doi: 10.1016/j.urology.2009.06.108. Epub 2009 Oct 24. PMID 19854483